CLINICAL TRIAL: NCT04204122
Title: Evaluation of Topical Vigamox in the Initial Management of Ocular Graft-Versus-Host Disease
Brief Title: Vigamox Treatment for Ocular Graft-Versus-Host Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decided to close study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202003066
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Ocular Graft-versus-host Disease
Keywords: GVHD; Graft-Versus-Host Disease; Ocular Surface; Ocular Surface Microbiome; Vigamox
MeSH Terms: conditions — Graft vs Host Disease | interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: The eyes of each enrolled participant will be randomized such that one eye is treated with Vigamox and the other eye is treated with a placebo eye drop.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Eye treated with Vigamox (Experimental): -The participant will be instructed to use one drop from each bottle four times per day for 7 days
  Interventions: Drug: Vigamox
- Arm 2: Eye treated with placebo (Placebo Comparator): -The participant will be instructed to use one drop from each bottle four times per day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vigamox — -FDA approved medication
  Other Names: Moxifloxacin
  Arms: Arm 1: Eye treated with Vigamox
Drug: Placebo — -The placebo is artificial tear drops
  Arms: Arm 2: Eye treated with placebo

SUMMARY:
In this study the investigators seek to prospectively measure the response of ocular graft-versus-host disease (GVHD) patients to treatment with topical Vigamox. The investigators will accomplish this by enrolling patients with bilateral ocular GVHD and treating one eye with topical Vigamox and the other eye with a placebo eye drop. By assessing the response to treatment with Vigamox, the investigators hope to identify a role for topical antibiotic treatment in ocular GVHD.

ELIGIBILITY:
Inclusion Criteria:

-Participants will be adults with a history of allogeneic hematopoietic stem cell transplantation, signs of either acute or chronic GVHD per the hematologist, signs and symptoms consistent with ocular GVHD + within 4 months of developing symptoms of ocular GVHD

Exclusion Criteria:

* Treated with antibiotic eye drops in the month prior to enrollment
* History of fluoroquinolone allergy
* Asymmetric ocular disease
* Pregnant
* Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Ocular comfort | First clinic visit through second clinic visit (estimated to be 9-14 days)
  * Ocular comfort will be rated by the participant for each eye on a 0-10 Visual Analog Scale
  * 0=no discomfort and 10=worst discomfort

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) score | First clinic visit through second clinic visit (estimated to be 9-14 days)
  * 12 questions with answers ranging from 0=none of the time to 4=all of the time
  * The OSDI©is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease.
Change in Visual acuity | First clinic visit through second clinic visit (estimated to be 9-14 days)
Change in the Degree of Conjunctival injection | First clinic visit through second clinic visit (estimated to be 9-14 days)
  -The degree of conjunctival injection will be graded based on the Validated Bulbar Redness scale
Change in Corneal/conjunctival punctate epithelial erosions | First clinic visit through second clinic visit (estimated to be 9-14 days)
  * The clinical exam will be conducted using the National Eye Institute Fluorescein Staining Scale to grade the degree of corneal and conjunctival stain with a cobalt blue slit lamp filter
  * This test divides the cornea into 5 sections. Staining is graded on a scale of 0-3, with 0 indicating absence of staining and 3 indicating severe staining.
Change in Culture results | First clinic visit through second clinic visit (estimated to be 9-14 days)
  -Conjunctival bacterial cultures will be obtained via swab before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Todd Margolis, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu